CLINICAL TRIAL: NCT03812757
Title: The Supraclavicular Fossa Ultrasound View for Correct Catheter Positioning in Infraclavicular Right Subclavian Central Venous Catheterization
Brief Title: Supraclavicular Fossa US View for Catheter Positioning in Right Subclavian Central Venous Catheterization
Status: Completed | Type: Observational
Sponsor: Skane University Hospital (Other)
Responsible Party: Principal Investigator, Ola Borgquist, Principal investigator, Skane University Hospital
Other Study IDs: CVC positioning
Record Dates: First submitted 2019-01-19; First posted 2019-01-23 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Central Venous Catheter Placement
Keywords: Central venous catheter; Subclavian vein; Supraclavicular fossa ultrasound view

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Supraclavicular fossa US scanning: Following insertion of at least 20 cm of the guidewire into the right subclavian vein, the probe is shifted to the right supraclavicular fossa to scan the right internal jugular vein in order to exclude malposition of the guidewire. The probe is then tilted in a caudal direction to obtain a view of the guidewire within the superior vena cava. Misplaced guidewires will be corrected under real-time ultrasound guidance.
  Interventions: Diagnostic Test: Supraclavicular fossa US scanning

INTERVENTIONS:
Diagnostic Test: Supraclavicular fossa US scanning — As previously stated.

SUMMARY:
The study will evaluate if the supraclavicular fossa ultrasound view can be used to achieve a correct catheter tip placement in infraclavicular right subclavian central venous catheter placement. This may make routine post-procedural x-ray exams redundant.

DETAILED DESCRIPTION:
Central venous catheterization is one of the most common procedures within intensive care medicine. Verification of correct catheter tip placement is a primary aspect of safety and quality of central venous catheterization as malposition may lead to life-threatening complications such as thrombosis, hemothorax, cardiac tamponade, and arrhythmias. Conventional chest x-ray (CXR) is routinely performed after every insertion and is considered gold standard to examine catheter tip location and evaluate for complications such as pneumo- and hemothorax. However, CXR exposes the patient to ionized radiation, requires a considerable amount of time, and is workload-generating for both ICU and radiology staff.

Weber et al has described the use of the right supraclavicular fossa view for real-time ultrasound-guided placement of a central venous catheter (CVC) via the right internal jugular vein (IJV) in adults. This approach has subsequently been validated in a clinical study and has also been used for supraclavicular subclavian line insertion. The approach requires use of a microconvex probe, which couples good image resolution and high scanning depth. The use of a microconvex probe for infraclavicular subclavian central venous catheter (CVC) insertion has been described previously, but this is the first description of the supraclavicular fossa ultrasound view to guide correct catheter tip placement in infraclavicular right subclavian CVC placement.

ELIGIBILITY:
Inclusion Criteria:

* Indication for central venous catheter placement.

Exclusion Criteria:

* Operator unable to visualize the subclavian vein (e.g., in those with subcutaneous emphysema of the chest wall),
* Subclavian vein catheterization deemed inappropriate by the operator,
* Central line/pacemaker/similar device already in place (risk for misinterpretation of the ultrasound image)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients >18 years with an indication for CVC placement and under the care of one of three intensivists responsible for the study will be consecutively included in the study
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Correct catheter tip positioning | Post-procedural x-ray (typically within 24 hours)
  Optimal placement (cavoatrial junction, distal superior vena cava); acceptable placement (upper part of the right atrium and entire SVC, provided that the axes of the catheter and vein are aligned to reduce the risk of vessel perforation); unacceptable placement (all other locations).

SECONDARY OUTCOMES:
Mechanical complications within 24 hours | Within 24 hours after central venous catheterization
  Bleeding, cardiac arrhythmias, arterial puncture/cannulation, pneumothorax.

CONTACTS AND LOCATIONS:
Overall Officials: Ola Borgquist, MD, PhD, Principal Investigator — Skane University Hospital
Locations (1):
- Skånes universitetssjukhus, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adrian M, Kander T, Lunden R, Borgquist O. The right supraclavicular fossa ultrasound view for correct catheter tip positioning in right subclavian vein catheterisation: a prospective observational study. Anaesthesia. 2022 Jan;77(1):66-72. doi: 10.1111/anae.15534. Epub 2021 Jul 14. PMID 34260061